CLINICAL TRIAL: NCT06031831
Title: Analysis of Epidemiology, Risk Factors, and Prognosis of Pediatric Patients After Operations for Congenital Heart Disease
Brief Title: Analysis of Risk Factors and Prognosis of Pediatric Patients After Operations for Congenital Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202205043RINB
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-05

CONDITIONS: Congenital Heart Disease; Pediatric
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: airway anomalies — with or without airway anomalies

SUMMARY:
This hospital-based retrospective study reviewed patients who underwent surgery for CHD between 2017 and 2020 and analyzed the clinical features and outcomes associated with airway anomalies.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric patients (age <18 years) who underwent surgery for CHD at our hospital between January 1, 2017, and December 31, 2020.

Exclusion Criteria:

* with much missing clinical data

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients (age <18 years) who underwent surgery for CHD at our hospital between January 1, 2017, and December 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 999 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
surgical mortality | 1 year
  hospital expired after operation
intermediate survival | 5 years
  expired during follow-up

SECONDARY OUTCOMES:
post-operative ICU stay | 1 year
  The length of ICU stay after operation
post-operative intubated days | 1 year
  The length of intubated days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Jenghung Wu, Taipei, Taiwan R., Taiwan

IPD SHARING:
Plan to Share IPD: Undecided